CLINICAL TRIAL: NCT06674486
Title: The Bio-equivalence Study of Iron Sucrose Injection in Healthy Participants
Brief Title: Bioequivalence Study of Iron Sucrose Injection in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sichuan Huiyu Pharmaceutical Co., Ltd (Industry)
Collaborators: Henan (Zhengzhou) Zhonghui Cardiovascular Hospital (Unknown); Changsha Duxact Biotechnology Co., Ltd (Unknown); Suzhou Guochen Biotechnology Co., Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: DUXACT-2409005
Record Dates: First submitted 2024-11-04; First posted 2024-11-05 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Bioequivalency; Safety Issues
MeSH Terms: interventions — Ferric Oxide, Saccharated; Long-Term Synaptic Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group I - Receive test product first and then reference product (Experimental)
  Interventions: Drug: Iron Sucrose injection (Test product, manufactured by Sichuan Huiyu Pharmaceutical Co., Ltd) and Iron Sucrose injection (Reference product, Venofer)
- Group II - Receive reference product first and then test product (Experimental)
  Interventions: Drug: Iron Sucrose injection (Reference product, Venofer) and Iron Sucrose injection (Test product, manufactured by Sichuan Huiyu Pharmaceutical Co., Ltd)

INTERVENTIONS:
Drug: Iron Sucrose injection (Test product, manufactured by Sichuan Huiyu Pharmaceutical Co., Ltd) and Iron Sucrose injection (Reference product, Venofer) — For the Group I, participants will receive a single intravenous injection of the Test Product (Iron sucrose injection, 100 mg iron/5 mL, manufactured by Sichuan Huiyu Pharmaceutical Co., Ltd). After a washout period, subjects will receive a single intravenous injection of the Reference Product (Iron sucrose injection, Venofer®, 100 mg iron/5 mL, held by Vifor France).
  Arms: Group I - Receive test product first and then reference product
Drug: Iron Sucrose injection (Reference product, Venofer) and Iron Sucrose injection (Test product, manufactured by Sichuan Huiyu Pharmaceutical Co., Ltd) — For the Group II, participants will receive a single intravenous injection of the Reference Product (Iron sucrose injection, Venofer®, 100 mg iron/5 mL, held by Vifor France) . After a washout period, subjects will receive a single intravenous injection of the Test Product (Iron sucrose injection, 100 mg iron/5 mL, manufactured by Sichuan Huiyu Pharmaceutical Co., Ltd).
  Arms: Group II - Receive reference product first and then test product

SUMMARY:
The goal of this clinical trial is to compare the pharmacokinetic profile of the single intravenous injection of the test product and reference product in healthy subjects and to evaluate the bio-equivalence and safety of these two injections in healthy subjects. The main questions it aims to answer are:

[Question 1] Is there significant difference in the pharmacokinetic profile between the Iron Sucrose Injection (100 mg/5 mL [calculated by iron]) manufactured by Sichuan Huiyu Pharmaceutical Co., Ltd. and the Iron Sucrose Injection (trade name: Venofer®, 100 mg/5 mL [calculated by iron]) held by Vifor France? [Question 2] Is it safe for the healthy subjects to take the test product (100 mg/5 mL [calculated by iron]) manufactured by Sichuan Huiyu Pharmaceutical Co., Ltd. and the reference product held by Vifor France? Participants will be randomly divided into group I and group II, with equal number of subjects in each group. Each subject will receive only one dose of either the test product or the reference product in each period (two-sequence crossover study).

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years, males or females;
2. Body weight ≥ 50.0 kg (male subjects) or ≥ 45.0 kg (female subjects), and body mass index (BMI) within 19-26 kg/m2 (both inclusive);
3. Subjects voluntarily sign a written informed consent form.

Exclusion Criteria:

1. Those who have a history of or currently have clinically serious diseases, including circulatory, endocrine, nervous, digestive, and respiratory, hematology, immunology, psychiatry and metabolic disorders or abnormalities or any other diseases that can interfere with the study results (e.g., non-iron deficiency anemia, history of severe asthma, hepatic or renal insufficiency);
2. Those with a history of iron deficiency or anemia within 6 months prior to the initial administration of the investigational drug;
3. Those with a history of allergy to two or more drugs (or foods), or allergy to iron, sucrose, or iron products;
4. Those who have undergone surgery within 28 days prior to the initial administration of the investigational drug, or who plan to undergo surgery during the study period;
5. Those who have been vaccinated within 28 days prior to the initial administration of the investigational drug, or who plan to be vaccinated during the study period;
6. Those who have received any medications or supplements (including herbal remedies) within 14 days prior to the initial administration of investigational drug;
7. Those who have used any iron supplements or iron-containing herbs or nutritional supplements within 3 months prior to the initial administration of the investigational drug;
8. Those who have used any drugs that inhibit or induce hepatic drug metabolism (e.g., inducers-barbiturates, carbamazepine, phenytoin and rifampicin; inhibitors-SSRIs, cimetidine, cyclosporine, macrolides, verapamil, quinolones, pyrrole-containing antifungals and HIV protease inhibitors) within 30 days prior to the initial administration of the investigational drug;
9. Those who have used any investigational medicinal product or been enrolled in any clinical studies of drugs/medical devices within 3 months prior to the initial administration of the investigational drug;
10. Those who have donated blood or had a blood loss volume of >400 mL within 3 months before the initial administration of the investigational drug;
11. Those who cannot tolerate venipuncture and/or have a history of hemophobia/fear of needles;
12. Those who have used oral contraceptives within 30 days before the initial administration of the investigational drug, or who have received long-acting estrogens or progesterone injections or implants within 6 months before the initial administration of the investigational drug;
13. Those (females) who have had unprotected sex within 14 days prior to the initial administration of the investigational drug, or females who are pregnant or breastfeeding;
14. Subjects and their partners who cannot take at least one non-medication contraceptive measures from signing the ICF to 3 months after the last administration, or those who plan to bear a child, or donate egg or sperm during this period;
15. Those who have special dietary requirements and are unable to comply with a uniform diet or have dysphagia;
16. Those who have consumed excessive amounts of tea, coffee or caffeinated beverages (more than 8 cups, 1 cup=250 mL) every day within 3 months prior to the initial administration of the investigational drug;
17. Those who have consumed or plan to consume any caffeine-containing foods/beverages (e.g., coffee, strong tea, chocolate) or foods (e.g., sardines, animal livers)/beverages that are rich in xanthine in the 48 h prior to the initial administration of the investigational drug;
18. Those who have consumed or plan to consume grapefruits or grapefruit-related citrus fruits (e.g., bigarades and pomelos), carambola, pawpaws and pomegranate, those who refuse to discontinue such diet during the study, or those who had strenuous exercises within 7 days prior to the initial administration of the investigational drug;
19. Those who are addicted to smoking or who have smoked no less than 5 cigarettes per day within 3 months prior to the initial administration of the investigational drug;
20. Those who are addicted to alcohol or who have frequently consumed alcohol, namely, consumed more than 14 units of alcohol every week (1 unit ≈ 200 mL of beer containing 5% alcohol, 25 mL of liquor containing 40% alcohol, or 85 mL of wine containing 12% alcohol) within 6 months prior to the initial administration of the investigational drug;
21. Those who abuse drugs or have used soft drugs (such as cannabis) within 3 months prior to the initial administration of the investigational drug, or have used hard drugs (such as morphine, methamphetamine, ketamine, THC, MDMA) within 1 year prior to the first use of the investigational drug;
22. Those with clinically significant abnormalities in vital signs, physical examination, 12-lead electrocardiogram, or laboratory tests as determined by the investigator, and those judged by the investigator to have increased safety risks if they continue to participate in the study;
23. Those who fail the alcohol test or are positive in the drug abuse screening upon admission;
24. Those who are unable to participate in the study due to their own reasons;
25. Those who are deemed unsuitable for participation in the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-11-22 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2025-03-14 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameter of total iron and transferrin-bound iron: Cmax | 36 hours, 24 hours, 12 hours and 0 hour before administration, 2, 6, 8, 10, 15, 30 and 45 minutes, 1, 2, 3, 4, 6, 8, 12, 14, 24, and 36 hours
  Cmax is the maximum observed concentration of total iron and transferrin-bound iron.
Pharmacokinetic parameter of total iron and transferrin-bound iron: AUC0-t | 36 hours, 24 hours, 12 hours and 0 hour before administration, 2, 6, 8, 10, 15, 30 and 45 minutes, 1, 2, 3, 4, 6, 8, 12, 14, 24, and 36 hours.
  AUC0-t is the area under the plasma concentration-time curve from time zero to time point t for the last measurable concentration of total iron and transferrin-bound iron.

CONTACTS AND LOCATIONS:
Locations (1):
- Henan (Zhengzhou) Zhonghui Cardiovascular Hospital, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No